CLINICAL TRIAL: NCT00540280
Title: Randomized Phase III Trial of Surgery Alone or Surgery Plus Preoperative Gemcitabine-Cisplatin in Clinical Early Stages of Non-small Cell Lung Cancer
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Follow up only
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Naeem Chaudhri, MD, King Faisal Specialist Hospital & Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAC#2031-059
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surgical Procedures, Operative

ARMS (1):
- Surgery alone (Active Comparator): Surgery alone
  Interventions: Radiation: Surgery alone or surgery plus preoperative Gemcitabine-Cisplatin

INTERVENTIONS:
Radiation: Surgery alone or surgery plus preoperative Gemcitabine-Cisplatin — Surgery + Chemo + RT

SUMMARY:
Randomized Phase III trial of surgery alone or surgery plus preoperative Gemcitabine-Cisplatin in clinical early stages of non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with early stage NSCLC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2003-10; Primary Completion 2003-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
OS, MS, DFS | overall

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Rehman, MD, Principal Investigator — King Faisal Specialist Hospital & Research Centre, Saudi Arabia